CLINICAL TRIAL: NCT06869369
Title: Pain Neuroscience Education for Middle School Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ismail Saracoglu, Head of Department, Kutahya Health Sciences University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: Turkish PNE4Kids
Record Dates: First submitted 2024-11-28; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Pain; Pediatrics; Neuroscience Pain Education; Physical Activity
Keywords: pain; pediatrics; neuroscience pain education; physical activity; sleep
MeSH Terms: conditions — Pain; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental)
  Interventions: Other: Turkish PNE4Kids
- control group (No Intervention)

INTERVENTIONS:
Other: Turkish PNE4Kids — Participants in the intervention group will receive 'Turkish PNE4Kids Programme'. The PNE4Kids program was developed based on the book "Explain pain" by Butler and Moseley and includes an explanation and reassurance on the cause of pain, a brief summary of relevant pain mechanisms, and the integral role of psychosocial and physical factors in precipitating and maintaining pain. This programme has been translated and validated in Turkish children.
  Arms: intervention group

SUMMARY:
This project was designed as a single-blind, randomised controlled, prospective intervention study. The research question of the project is 'Is pain neuroscience education an effective method to improve various aspects of child health, conceptualise pain and change pain-related behaviours in middle school children?'. In other words, the aim of this project is to investigate whether pain neuroscience education (PNE4Kids) is an effective method for improving various aspects of child health, conceptualising pain and changing pain-related behaviours in middle school children. For this purpose, it is planned to implement PNE4Kids based power point presentation and interactive game training. It is aimed to evaluate children in terms of physical activity level, sleep quality/habits, pain conceptualisation level and participation in leisure time activities. Physical activity levels will be assessed with Actigraph GT3X+ accelerometer device and 'Physical Activity Scale for Older Children'. Sleep quality/ habits will be assessed with Actigraph GT3X+ accelerometer and 'Children's Sleep Habits Scale-short form'. Knowledge of pain conceptualisation will be assessed with the 'Conceptualisation of Pain' scale. Children's level of participation in leisure time activities will be assessed through the participation section/domain of the Participation Environment Measure for Children and Youth (PEM-CY). After the baseline measurements of the individuals included in the study and who volunteered will be completed, they will be randomly assigned to the control or intervention group. Participants in the intervention group will receive 'Turkish PNE4Kids Programme'. Individuals in the control group will not receive any intervention. All evaluations will be repeated before the training, immediately after the training and at the end of the 3rd month after the training.

ELIGIBILITY:
Inclusion Criteria:

* Being actively educated at midschool level,
* Having sufficient reading and understanding skills in Turkish.

Exclusion Criteria:

* Chronic pain (pain in ≥1 anatomic region that persists or recurs for longer than 3 months,
* Chronic illness (e.g. cancer, diabetes, asthma, juvenile rheumatic arthritis),
* Being diagnosed with a specific learning disability,
* Being diagnosed with attention deficit hyperactivity disorder,
* Being diagnosed with autism spectrum disorder,
* Not being willing to participate in the study by oneself or one's parents.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 57 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Physical Activity Level | Change from Baseline at 3 months
  Children's physical activity levels will be assessed with the "Physical Activity Questionnaire for Older Children (PAQ-C 8-14)". The scale is an assessment tool that children can self-administer, developed by Crocker et al (Crocker et al., 1997) for children in the 4th to 8th grades. There is also a form of the same scale developed for adolescents (Kowalski et al., 1997). The physical activity scale developed for older children has a total of 10 items based on a 5-point Likert scale (1 point: lowest, 5 points: highest) that measure children's physical activity levels in the last week.
Sleep Quality | Change from Baseline at 3 months
  In order to evaluate children's sleep prices, the Child Sleep Habits Questionnaire-short formulas, which were separated by Owens and colleagues (Owens et al., 2000) in 2000 and comprehensively covering children's sleep quality and sleep conduction, will be used (Owens et al., 2000). The questionnaire, which can be done in Turkish and has been made reliable by Balık et al. (Fis et al., 2011), consists of a total of 33 items. The total score of 41 is accepted as the cut-off point and values above this are evaluated as 'clinically significant sleep disturbance'.
Pain conceptualization/knowledge level | Change from Baseline at 3 months
  Children's pain concept (pain knowledge, beliefs and attitudes towards pain) levels will be assessed with the "Pain Conceptualization Scale (COPI)".
  The Pain Conceptualization Scale is a 14-item scale developed by Pate et al (Pate et al., 2020) to assess children's pain knowledge, beliefs and attitudes towards pain. This scale includes pain-related items based on 7 areas suggested by pediatric pain specialists. Each item is evaluated according to a 5-point Likert Scale ranging from "strongly agree (4 points)" to "strongly disagree (0 points)".
  Higher scores indicate higher levels of compliance with pain science.
Leisure Time/Activity Participation | Change from Baseline at 3 months
  Children's participation in leisure activities will be assessed through the participation section/domain of the Participation Environment Measure for Children and Youth (PEM-CY) (Coster et al., 2011). The participation section in the PEM-CY consists of 10 items for home environments, 5 items for school environments, and 10 items for community environments. This scale will be administered by the children's parents.

SECONDARY OUTCOMES:
School attandence level | Change from Baseline at 3 months
  Children's school attendance will be evaluated with the "e-school absence tracking" (Golcuk, 2015) system. This information will be requested from the school administration. Beforehand, parents will be contacted by phone and their consent will be obtained with the Personal Data Protection (PDPL) Informed Consent Form.
Physical education class attendance level | Change from Baseline at 3 months
  This information will be requested from physical education teachers. Parents will be contacted by phone beforehand and their consent will be obtained with the Personal Data Protection (PDP) Informed Consent Form. Children's attendance to physical education classes will be evaluated by the physical education teacher by answering the following questions:
  • Has he/she missed physical education classes due to pain in the last 3 months - yes/no; if yes, how many days/lessons?
Doctor/hospital visits | Change from Baseline at 3 months
  Information on the frequency of children's doctor visits will be requested from the children's parents. The parents will be contacted by phone and their consent will be obtained with the Informed Consent Form on the Protection of Personal Data (KVK) beforehand.
  Question 1: How many times have you been to the doctor in the last 3 months because you had pain somewhere?
  1. We never did.
  2. We went once
  3. We went more than once.
  Question 2: Have you received rehabilitation treatment (physical therapy, exercise, manual therapy, etc.) in the last 3 months because you had pain somewhere?
  1. We never did.
  2. We did once.
  3. We did more than once.
Using of pain killers | Change from Baseline at 3 months
  Information on the frequency of children's medication use will be requested from the children's parents. The parents will be contacted by phone and their consent will be obtained with the Informed Consent Form on the Protection of Personal Data (KVK) beforehand.
  Question 1: How many times have I used medication in the last 3 months because I had pain somewhere?
  1. We never did.
  2. We used once.
  3. We used more than once.

CONTACTS AND LOCATIONS:
Overall Officials: Esra AKIN, Ph.D., Principal Investigator — Kutahya Health Sciences University; İnci ARIKAN, Prof. Dr., Principal Investigator — Kutahya Health Sciences University; Kelly ICKMANS, Ph.D., Principal Investigator — Vrije Universiteit Brussels; Emma RHEEL, Ph.D., Principal Investigator — Vrije Universiteit Brussels
Locations (1):
- Kutahya National Education Directorate, Kütahya, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kara OK, Gursen C, Ickmans K, Rheel E, Elma O, Cetin SY, Dogan M, Kutluk MG, Kara K. Enhancing pediatric pain management in Turkey: A modified Delphi study on culturally adapted pain neuroscience education for chronic pain in children. J Pediatr Nurs. 2024 Nov-Dec;79:91-99. doi: 10.1016/j.pedn.2024.09.001. Epub 2024 Sep 7. PMID 39243665
- [Background] Pas R, Meeus M, Malfliet A, Baert I, Oosterwijck SV, Leysen L, Nijs J, Ickmans K. Development and feasibility testing of a Pain Neuroscience Education program for children with chronic pain: treatment protocol. Braz J Phys Ther. 2018 May-Jun;22(3):248-253. doi: 10.1016/j.bjpt.2018.02.004. Epub 2018 Mar 4. PMID 29550259